CLINICAL TRIAL: NCT03138837
Title: Role of 3 Tesla Diffusion Weighted Magnetic Resonance Imaging (DW-MRI) for Diagnosis Bladder Cancer Grade and Stage. Potential Role of the Apparent Diffusion Coefficient (ADC) Value
Brief Title: Role of 3 Tesla Diffusion Weighted Magnetic Resonance Imaging (DW-MRI) for Diagnosis Bladder Cancer Grade and Stage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Other Study IDs: R/17.02.31
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Diagnoses Disease; Magnetic Resonance Imaging; Apparent Diffusion Coefficient
Keywords: Bladder cancer; Magnetic Resonance Imaging; Bladder Cancer Superficial
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder Biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Diffusion Weighted Magnetic resonance imaging

SUMMARY:
assess diagnostic performance of 3-Tesla DW-MRI in detecting and staging bladder cancer and potential role of the ADC value as a biomarker reflecting histological grade and stage.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older
* Suspected by the out-patient flexible cystoscopy as Non-muscle invasive bladder cancer.
* Patient who will undergo radical cystectomy.
* Patient with history of allergy to iodinated contrast media

Exclusion Criteria:

* Refuse to complete study requirements
* Patient with any of the following:

  1. Any metallic fragment or foreign body
  2. Coronary and peripheral artery stents
  3. Aortic stent graft
  4. Prosthetic heart valves and annuloplasty rings
  5. Cardiac pacemaker
  6. Implanted cardioverter-defibrillator (ICD)
  7. Retained trans venous pacemaker and defibrillator leads
  8. Cochlear, otologic, or other ear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of participants from single tertiary centre outpatient clinic of Urology and Nephrology Center in Mansoura
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
assess the diagnostic performance of 3-T DW-MRI in detecting and staging bladder cancer | 1 year
  comparing the radiological diagnosis with the pathological specimen results

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abol-Enein, MD, Study Chair — Urology and Nephrology center; Mohamed AboElghar, MD, Study Director — Urology and Nephrology center; Ahmed O. Mosbah, MD, Principal Investigator — Urology and Nephrology center; Khaled Sheir, MD, Principal Investigator — Urology and Nephrology center; Ahmed Elassmy, MD, Principal Investigator — Urology and Nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Hassan Abol-Enein, MD, Phd (Study Chair)